CLINICAL TRIAL: NCT05869331
Title: Midterm (Min. 3yr) Follow-up of Patients With Single Spiral/Oblique Finger Metacarpal Fracture Following Early Mobilization Nonoperative Treatment or Operative Treatment With Screw Fixation - a Noninferiority Randomized Controlled Trial
Brief Title: Midterm (Min. 3yr) Follow-up of Patients With Single Spiral/Oblique Finger Metacarpal Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 276742
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Metacarpal Fracture
Keywords: Metacarpal fracture; Spiral fracture; Early mobilization
MeSH Terms: conditions — Fractures, Bone | interventions — Early Ambulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nonoperative treatment (Experimental): Patients in this group were treated with early mobilization.
  Interventions: Procedure: Early mobilization
- Operative treatment (Active Comparator): Patients in this group were treated surgically.
  Interventions: Procedure: Operative treatment

INTERVENTIONS:
Procedure: Early mobilization — Patients randomized to nonoperative treatment have already received treatment using early mobilization in the original trial, and all fractures have been confirmed healed. Mobilization consisted of 5 repetitions of full finger extension followed by maximum finger flexion, and 5 such sets of 5 were required per day for the first 6 weeks. Buddy taping or resting splint was offered if the patient experienced difficulty, and mobilization was performed by all patients in this treatment arm.
  Arms: Nonoperative treatment
Procedure: Operative treatment — Patients randomized to operative treatment have already received treatment using open reduction and internal fixation (ORIF) with cortical screws in the original trial, and all fractures have been confirmed healed. Surgery was performed under general anaesthesia through a dorsal incision centered over the fractured metacarpal. Reduction was performed under visual inspection and fixation performed using 2 or more cortical screws (Synthes Compact Hand 2.0) as first option. At the surgeons preference fixation using plate and screw fixation was also allowed. Postoperatively patients were put in a plaster cast for two weeks and then hand therapy was initiated.
  Arms: Operative treatment

SUMMARY:
Spiral metacarpal fractures (metacarpal II-V) can be treated conservatively or with operation. With minimal displacement this fracture is usually treated with immobilisation or early mobilisation. With appreciable displacement especially any malrotation the patient usually is treated with an operation. This usually includes an open reduction of the fracture and fixation with plates and screws or just screws.

The hypothesis that nonoperative treatment (using early mobilization without splintage) will result in similar outcomes to operative treatment was previously tested by this research group (Peyronson et al. JBJS American 2023). Over a 1-year follow-up the primary outcome of grip strength was found to be noninferior.

This trial will extend the follow-up period and re-evaluate the patients included in the original cohort to identify any difference over a 3-6 year follow up.

DETAILED DESCRIPTION:
The original trial was a noninferiority randomized controlled trial evaluating 42 patients. Randomization was performed 1:1 to either nonoperative treatment with mobilization initiated immediately following recruitment or operative treatment using ORIF with cortical screws or locking compression plate (LCP) and screw fixation.

The non-inferiority margin (NIM) was defined as -15% grip strength of the injured hand relative to the contralateral hand. The same NIM will be used for this trial.

Because subtle biomechanical changes (mainly metacarpal bone shortening) could theoretically cause problems not evident at 1-year follow-up (such as joint degeneration from changes in load distribution), the investigators plan to re-evaluate the patients for a longer-term follow-up.

Only patients included in the original trial will be eligible for inclusion in this extended follow-up. Participation will be offered via mail invitation, and participants will be offered financial compensation in the form of a single payment of 500SEK.

Data collection will be performed in a single outpatient hospital visit where patient history, subjective outcome data and bilateral plain radiography of the hands will be obtained.

ELIGIBILITY:
Inclusion Criteria:

Previous inclusion in the original study population, i.e.:

* Diaphyseal, single spiral, and oblique fractures of the index to little finger metacarpals
* Fracture line length at least twice the diameter of the bone at the level of the fracture
* At least 2-mm displacement and/or shortening of the fracture or malrotation
* Normal hand function before the injury
* Fracture <10 days old

Exclusion Criteria:

* Multiple metacarpal fractures
* Open fractures
* Inability to follow instructions
* Fracture line length less than twice the diameter of the bone at the level of the fracture
* Abnormal hand function before the injury
* Previous ipsilateral hand fractures
* Fracture ≥10 days old at possible randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Grip strength | 3-6 years
  Grip strength is measured in both hands using a JAMAR dynamometer set to 2nd position with the patient sitting down, arm resting in 90 degree elbow flexion and neutral forearm rotation. Three measurements are taken in each arm and the mean value calculated. The strength of the injured hand is expressed as a percentage value relative to the strength of the contralateral (uninjured) hand.

SECONDARY OUTCOMES:
DASH score | 3-6 years
  Disability of Arm, Shoulder and Hand questionnaire score, a patient-reported outcome measure. Scored 1-100, 1 representing best possible value.
Metacarpal shortening | 3-6 years
  Shortening of the metacarpal bone measured on plain radiographs comparing the length of the injured bone to the contralateral corresponding bone and calculating the difference in millimeters.
Rotation | 3-6 years
  Presence of any rotation deformity on clinical examination
Subjective pain | 3-6 years
  Pain graded by patient using a numeric rating scale (NRS) 1-10, 1 representing best possible value
Subjective cosmetic result | 3-6 years
  Cosmetic result graded by patient using a numeric rating scale (NRS) 1-10, 1 representing best possible value
Subjective overall result | 3-6 years
  Overall result of treatment outcome graded by patient using a numeric rating scale (NRS) 1-10, 1 representing best possible value
Time off work | 3-6 years
  The time off work measured in days, or time until return to normal function (in retired patients or patients attending education)
Range of motion | 3-6 years
  Range of motion of the affected finger ray presented as total active motion (TAM)

CONTACTS AND LOCATIONS:
Overall Officials: Björn Äng, Professor, Study Chair — Region Dalarna
Locations (2):
- Sweden (2):
  - Falun Regional Hospital, Falun
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peyronson F, Ostwald CS, Hailer NP, Giddins G, Vedung T, Muder D. Nonoperative Versus Operative Treatment for Displaced Finger Metacarpal Shaft Fractures: A Prospective, Noninferiority, Randomized Controlled Trial. J Bone Joint Surg Am. 2023 Jan 18;105(2):98-106. doi: 10.2106/JBJS.22.00573. Epub 2022 Nov 10. PMID 36455163